CLINICAL TRIAL: NCT00516087
Title: Administration of LMP1- and LMP2-Specific Cytotoxic T-Lymphocytes to Patients With EBV-Positive Nasopharyngeal Carcinoma
Brief Title: LMP1- and LMP2-Specific CTLs to Patients With EBV-Positive NPC (NATELLA)
Acronym: NATELLA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other); Center for Cell and Gene Therapy, Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Stephen Gottschalk, Associate Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21000-NATELLA; NATELLA; NCT00682864 (obsolete NCT alias)
Record Dates: First submitted 2007-08-10; First posted 2007-08-14 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Patients (Experimental): Patients with NPC in first or subsequent relapse or with primary refractory disease or high risk (T3 or T4, or node positive disease) in whom the EBV genome or antigens have been demonstrated in tissue biopsies.
  Interventions: Biological: Genetically modified CTLs

INTERVENTIONS:
Biological: Genetically modified CTLs — LMP1- and LMP2-specific T cells will be given by intravenous injection over 1-10 minutes through either a peripheral or a central line.
  Three different dosing schedules will be evaluated. Each patient will receive two injections, 14 days apart, according to the following dosing schedules:
  Group One Day 0 2x10^7 cells/m2 Day 14 2x10^7 cells/m2
  Group Two Day 0 2x10^7 cells/m2 Day 14 1x10^8 cells/m2
  Group Three Day 0 1x10^8 cells/m2 Day 14 2x10^8 cells/m2

SUMMARY:
Patients have a type of cancer called nasopharyngeal carcinoma (NPC) which has either come back, not gone away or is at high risk for coming back after the best treatment we know for this disease. We are inviting patients to participate in a research study using a new experimental therapy consisting of special immune system cells called LMP1- and LMP2-specific cytotoxic T lymphocytes (LMP1- and LMP2-CTLs).

Some patients with nasopharyngeal carcinoma show evidence of infection with the virus that causes infectious mononucleosis Epstein Barr virus (EBV) before or at the time of their diagnosis. EBV is found in the cancer cells of almost all patients with advanced stage NPC, suggesting that it may play a role in causing the disease. The cancer cells infected by EBV are able to hide from the body's immune system and escape destruction. We want to see if special white blood cells, called T cells, that have been trained to recognize and kill special parts of EBV infected cells can survive in blood and affect the tumor.

We have used this sort of therapy to treat a different type of cancer that occurs after bone marrow and solid organ transplant called post-transplant lymphoma. In this type of cancer the tumor cells have 9 proteins made by EBV on their surface. We grew T cells in the laboratory that recognized all 9 proteins and were able to prevent and treat post-transplant lymphoma. However nasopharyngeal carcinoma tumor cells only express 2 EBV proteins (LMP1 and LMP2) on their surfaces. In a previous study we made T cells that recognized all 9 proteins and gave them to patients with NPC. While some patients had a response, only a few patients had their cancer completely go away. We are now trying to find out if we can improve this treatment by growing and giving T cells where more of the cells will recognize two of the proteins expressed on NPC cells called LMP1 and LMP2. These special T cells are called LMP1- and LMP2-CTLs. These LMP1- and LMP2-CTLs are an investigational product not approved by the Food and Drug Administration.

DETAILED DESCRIPTION:
Patients have an EBV-positive cancer. We had gotten permission to take blood from patients in the past, which was used to grow T cells in the laboratory. We first grew a special type of cell called dendritic cells to stimulate the T cells. We then put a specially produced human virus (adenovirus) that carries the LMP1 and LMP2 gene into the dendritic cells. These dendritic cells were then treated with radiation so they could not grow. They were then used to stimulate T cells. This stimulation trained the T cells to kill cells with LMP1 and LMP2 on their surface. We then grew these LMP1- and LMP2-specific CTLs by more stimulation with EBV infected cells (which we made from blood by infecting them with EBV in the laboratory and treated them with radiation so they would not grow). We also put the adenovirus that carries the LMP1 and LMP2 genes into these EBV infected cells so that we increase the amount of LMP1 and LMP2 that these cells have. Once we made sufficient numbers of T cells we tested them to make sure they kill cells with LMP1 and LMP2 on their surface. These cells are now ready to give to the patients if they agree to participate in this study.

If the patient agrees to this treatment they will get treated with two doses of LMP1-and LMP2-specific CTLs, each dose given 2 weeks apart. If the patient is a female of child-bearing potential, we will give them a pregnancy test within one week prior to the infusion. If the patient is pregnant, they will not be able to participate in the study. The study doctor will be notified.

The CTLs will be thawed and injected through a central line, if they have one, or through a vein in their arm over 1 to 10 minutes. They may receive a dose of Tylenol and Benadryl beforehand. We will then monitor the patient in clinic for 1 to 4 hours after the injection.

All of the treatments will be given by the Center for Cell and Gene Therapy at Texas Children's Hospital or Houston Methodist Hospital. We will follow the patient in the clinic after the CTL injection and also follow results of their disease evaluations with the primary doctor.

To learn more about the way the T cells are working and how long they last in the body, an extra 10-60 mls (2-12 teaspoonfuls) of blood will be taken. We will use this blood to look at the immune response in the blood to the cancer.

To learn if the injected T cells have anti-tumor activity, we will measure the size of the patient's tumor before the T-cell infusion and 8 weeks afterwards with routine imaging studies such as CT (computer tomogram), MRI (magnetic resonance imaging), or PET (Positron Emission Tomography). If the patient has stable disease or there is a reduction in the size of the tumor on imaging studies after the T-cell infusion, the patient can receive up to six additional doses of the T cells at 6 to 12 weeks intervals if they wish.

ELIGIBILITY:
Inclusion Criteria:

All patients with NPC in first or subsequent relapse or with primary refractory disease or high risk (T3 or T4, or node positive disease) in whom the EBV genome or antigens have been demonstrated in tissue biopsies will be eligible for this trial.

Any patient with EBV positive NPC, in relapse or with primary resistant disease

Patients with a life expectancy 6 weeks or greater

Patients with bilirubin less than 2x normal, SGOT less than 3x normal, and Hgb more than 8.0.

Patients with a Karnofsky score (age greater than/=16) of or Lansky score (age less than 16) of greater than/= 50

Patients with a creatinine 2x normal for age or less

Patients should have been off other investigational therapy for one month prior to entry in this study

Patient, parent/guardian able to give informed consent

Exclusion Criteria:

Severe intercurrent infection

Due to unknown effects of this therapy on a fetus, pregnant women are excluded from this research. The male partner should use a condom.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2007-08; Primary Completion 2012-12 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
adverse events are being measured/assessed for the safety of autologous LMP1- and LMP2- specific cytotoxic T-lymphocytes (CTL) in patients with EBV-positive nasopharyngeal carcinoma (NPC). | 12 months

SECONDARY OUTCOMES:
Adverse events will be measured/obtained for information on the expansion, persistence and anti-tumor effects of autologous LMP1- and LMP2 specific CTL in patients with EBV-positive NPC. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Gottschalk, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Houston Methodist Hospital, Houston, Texas
  - Texas Children's Hospital, Houston, Texas